CLINICAL TRIAL: NCT03551275
Title: A Multicenter Open-Label Non-Comparative Dose Escalation Study (Phase 1) of the Pharmacodynamics, Pharmacokinetics, Safety, and Immunogenicity of BCD-132 (JSC BIOCAD, Russia) in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Dose Escalation Study of the Pharmacodynamics, Pharmacokinetics, Safety, and Immunogenicity of BCD-132 in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: BCD-132-1
Record Dates: First submitted 2018-02-13; First posted 2018-06-11 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: BCD-132; Multiple Sclerosis; anti-CD20
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort no. 1, BCD-132, 100 mg, IV (Experimental): Cohort no. 1, Group #1 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 100 mg.
  Cohort no. 1, Group #2 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 50 mg and second dose of 50 mg IV after 14 days period after first infusion.
  If there is no DLT within the first 14 days after infusion then Cohort no.2 is included.
  Interventions: Biological: BCD-132
- Cohort no. 2, BCD-132, 250 mg, IV (Experimental): Cohort no. 2, Group #3 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 250 mg.
  Cohort no. 2, Group #4 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 125 mg and second dose of 125 mg IV after 14 days period after first infusion.
  If there is no DLT within the first 14 days after infusion then Cohort no.3 is included.
  Interventions: Biological: BCD-132
- Cohort no. 3, BCD-132, 500 mg, IV (Experimental): Cohort no. 3, Group #5 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 500 mg.
  Cohort no. 3, Group #6 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 250 mg and second dose of 250 mg IV after 14 days period after first infusion.
  If there is no DLT within the first 14 days after infusion then Cohort no.4 is included.
  Interventions: Biological: BCD-132
- Cohort no. 4, BCD-132, 1000 mg, IV (Experimental): Cohort no. 4, Group #7 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 1000 mg.
  Cohort no. 4, Group #8 includes 3 (+3) subjects who will receive the single intravenous infusion of BCD-132 at the dose of 500 mg and second dose of 500 mg IV after 14 days period after first infusion.
  Interventions: Biological: BCD-132

INTERVENTIONS:
Biological: BCD-132 — Dose Escalation Study
  Other Names: humanized monoclonal antibody against CD20

SUMMARY:
BCD-132 is a humanized monoclonal antibody against CD20. BCD-132-1 is a Multicenter Open-Label Non-Comparative Dose Escalation Study (Phase 1) of the Pharmacodynamics, Pharmacokinetics, Safety, and Immunogenicity of BCD-132 (JSC BIOCAD, Russia) in Patients with Relapsing-Remitting Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent to participate in the study;
* Men and women aged from 18 to 60 years (inclusive) on the day of signing informed consent;
* Confirmed diagnosis of relapsing-remitting multiple sclerosis (according to McDonald criteria 2010);
* Documentary evidence that within the last 12 months before signing informed consent the patient had:

  1. At least one relapse, or
  2. At least one gadolinium enhancing T1-weighted lesion or one new T2-weighted lesion in dynamics.
* The patient should be neurologically stable during 30 days before signing informed consent (i.e. the patient should not have any new or aggravated neurological symptoms during this period, as told by the patient; or the patient's condition should be completely stabilized since the last relapse, and the duration of stabilization should be at least 30 days);
* A total EDSS score of 0 to 5.5 inclusive (assessed by the Assessing Neurologist);
* Presence of IgG antibodies to varicella zoster virus according to screening results;
* Patients of childbearing potential and their partners with preserved reproductive function must implement reliable contraceptive methods starting from signing informed consent and throughout the study. This requirement does not apply to patients after operative sterilization. Reliable contraception methods include one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives.
* Body weight ≥65 kg at the screening
* The absence of suicidal ideation and suicidal behavior, as assessed by the C-SSRC scale, for the period of the 1st month preceding the signing of the informed consent by the patient (0 score in the evaluation of suicidal ideation and the lack of positive responses in the section of suicidal behavior) established in the screening.

Exclusion Criteria:

* Primary and secondary progressive multiple sclerosis;
* Multiple sclerosis duration of more than 10 years with EDSS score ≤2.0 according to screening results;
* Other conditions (except for multiple sclerosis) that can affect the assessment of multiple sclerosis symptoms: to mask, aggravate, change symptoms of multiple sclerosis, result in clinical signs or laboratory instrumental findings suggesting multiple sclerosis;
* A relapse during the screening period;
* Any acute infections, relapses of chronic infections or any other chronic diseases that are present on the day of signing informed consent and can, as judged by the Investigator, negatively affect the patient's safety during the study treatment;
* HIV, hepatitis B, hepatitis C, or syphilis;
* Metabolic abnormalities (disorders) manifesting as:

  1. baseline creatinine levels increased more than 2-fold vs. upper limit of normal;
  2. baseline urea levels increased more than 3-fold vs. upper limit of normal;
  3. baseline ALT, AST or GGT levels increased more than 2.5-fold vs. upper limit of normal;
  4. baseline bilirubin levels increased more than 1.5-fold vs. upper limit of normal;
* Baseline leukocyte counts lower than <3.0 × 10 9/L, platelet counts lower than <125 × 10 9/L or hemoglobin levels <100 g/L;
* A history of severe depression, suicidal thoughts or suicide attempts;
* Signs of clinical significant depression (baseline Beck's score of more than 15);
* A history of hypothyroidism/hyperthyroidism and/or baseline abnormalities of TSH levels vs. lower or upper limits of normal;
* Epilepsy;
* Pregnancy, lactation or planned pregnancy over the entire study period;
* A history of use

  1. any time before signing informed consent: anti-B-cell agents (e.g., rituximab, ocrelizumab, abatacept, belimumab, ofatumumab, etc.);
  2. any time before signing informed consent: alemtuzumab, anti-CD4 agents, daclizumab, teriflunomide, laquinimod, mitoxantrone, cladribine, total lymphatic irradiation, bone marrow transplant;
  3. within 2 years (24 months) before signing informed consent: cyclophosphamide, cyclosporin, azathioprine; mycophenolate mofetil, fingolimod and other sphingosine-1-phosphate (S1P) receptor-modulating agents, natalizumab ;
  4. therapy with immunoglobulin drug products within 12 weeks before signing informed consent.
* Systemic corticosteroids used within 30 days before signing informed consent;
* Hypersensitivity to any of BCD-132 ingredients;
* Known alcoholic or drug dependency or signs of present alcoholic/drug dependence that, in the Investigator's opinion, can be contraindications for study therapy of multiple sclerosis with anti-CD20 monoclonal antibodies or limit treatment compliance;
* Inability to follow the Protocol procedures (in the Investigator's opinion);
* Contraindications to MRI or use of gadolinium-containing contrast agents:

  1. Metal foreign objects in the body, magnetic implants, ferromagnetic clips for cerebral vessels, artificial heart valves, electronic middle ear implants, pacemakers;
  2. A history of allergy to gadolinium or gadolinium-containing contrast agents;

  с) Fear of cramped spaces; d) Kidney function impairment with a risk of delayed gadolinium elimination (creatinine level increased to more than 2 x upper limit of normal); e) Documented diagnosis of sickle cell or hemolytic anemia, hemoglobinopathy.
* Any malignancies or a history of malignancies, except for cured basal cell carcinoma or cervical cancer in situ;
* Vaccination within 6 weeks before signing informed consent (as told by the patient);
* Participation in other clinical studies within 90 days before signing informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who developed AEs/SAEs that, in the Investigator's opinion, are related to BCD-132 | day 169
The proportion of patients, in each group, who developed СТСАЕ v. 4.03 Grade 3-4 AEs that, in the Investigator's opinion, are related to BCD-132 | day 169
The proportion of patients, in each group, who discontinued the study due to AEs/SAEs | day 169
The proportion of BAb- and NAb-positive patients | day 169

SECONDARY OUTCOMES:
AUC (0-2016 hours) | day 85, day 169
AUC (0-∞) | day 85, day 169
AUEC (0-2016 hours) | day 85, day 169
AUEC (0-∞) | day 85, day 169

OTHER OUTCOMES:
CUA | day 169
  Changes in MRI markers
Proportion of patients without contrast-enhancing lesions | day 169
  Changes in MRI markers
Number of new or enlarging T2-weighted lesions | day 169
  Changes in MRI markers over time
Proportion of patients without new or enlarging T2-weighted lesions | day 169
  Changes in MRI markers
Changes in T2-weighted lesion volume | day 169
  Changes in MRI markers
Changes in hypointense T1-weighted lesion volume | day 169
  Changes in MRI markers
Expanded Disability Status Scale (EDSS) | day 169
  EDSS is a scale for assessing neurologic impairment in MS. It consists of eight functional systems (FS) which are used to derive the EDSS steps (score) ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's score is determined between 0 to 10. A positive change from baseline indicates improvement
Proportion of relapse-free patients | day 169

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - City Hospital #15, Moscow
  - Moscow Regional Research and Clinical Institute, Moscow
  - Scientific Center of Neurology, Moscow
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Institute of the Human Brain n. a. N.P. Bekhtereva Russian Academy of Sciences, Saint Petersburg